CLINICAL TRIAL: NCT05704361
Title: A Multiple-center, Non-randomized, Open-label, Adaptive, Single-ascending Dose (Part 1 and Part 2) and Multiple-ascending Dose (Part 3) Parallel, Phase IB Study to Investigate the Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of RO7121932 Following Intravenous (Parts 1) and Subcutaneous Administration (Parts 2 and 3) in Participants With Multiple Sclerosis
Brief Title: A Study to Investigate the Safety, Tolerability, and Processing by the Body of Intravenous and Subcutaneous RO7121932 Administration in Participants With Multiple Sclerosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP42230; 2020-004122-33 (EudraCT Number); 2023-509357-31-00 (EU CTIS Number)
Record Dates: First submitted 2023-01-04; First posted 2023-01-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Single Ascending Dose (SAD) IV: RO7121932- Dose Escalation Cohorts 1 to 6 and Later Cohorts (Experimental): Participants will receive a single IV dose of RO7121932 on treatment Day 1. The planned starting dose of RO7121932 is 7 milligrams (mg) and will be escalated up to 2000 mg. The maximum dose will not exceed 4000 mg . Doses may be repeated, adjusted downwards, or intermediate doses may be investigated based on emerging data.
  Interventions: Drug: RO7121932 IV
- Part 2: SAD SC: RO7121932- Dose Escalation Cohorts 1 to 2 (Experimental): Participants will receive a single SC dose of RO7121932 on treatment Day 1. The planned starting dose of RO7121932 is 70 mg and will be escalated up to 200 mg. Doses may be repeated, adjusted downwards, or intermediate doses may be investigated based on emerging data.
  Interventions: Drug: RO7121932 SC
- Part 3: Multiple Ascending Dose (MAD) SC: RO7121932- Dose Escalation Cohorts 1 to 3 (Experimental): Participants will receive multiple SC doses of RO7121932, once weekly on treatment Day 1 through Day 22. The planned starting dose of RO7121932 is 70 mg and will be escalated up to 700 mg. Doses may be repeated, adjusted downwards, or intermediate doses may be investigated based on emerging data.
  Interventions: Drug: RO7121932 SC

INTERVENTIONS:
Drug: RO7121932 IV — Participants will receive RO7121932, as an IV infusion, per the schedule specified in the treatment arms.
  Arms: Part 1: Single Ascending Dose (SAD) IV: RO7121932- Dose Escalation Cohorts 1 to 6 and Later Cohorts
Drug: RO7121932 SC — Participants will receive RO7121932, as SC injection, per the schedule specified in the treatment arms.
  Arms: Part 2: SAD SC: RO7121932- Dose Escalation Cohorts 1 to 2; Part 3: Multiple Ascending Dose (MAD) SC: RO7121932- Dose Escalation Cohorts 1 to 3

SUMMARY:
The primary purpose of the study is to evaluate the safety and tolerability of a single-ascending intravenous (IV) dose (Part 1), a single-ascending subcutaneous (SC) dose (Part 2), and multiple ascending SC doses (Part 3) of RO7121932 in participants with multiple sclerosis (MS).

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Scale (EDSS) score ≤7.0 at Screening
* Participants with relapsing multiple sclerosis (RMS) or progressive multiple sclerosis (PMS) who fulfil international panel criteria for diagnosis (McDonald 2017 criteria)
* Participants not treated with any approved MS treatment at Screening and not planning to start on any MS therapy during the study (including follow-up)
* Female participants must practice abstinence or otherwise use contraception

Exclusion Criteria:

* Evidence of clinical disease activity as defined by any clinical relapse within 3 months prior to screening, or by >1 clinical relapse within 12 months prior to screening
* Evidence of magnetic resonance imaging (MRI) activity as defined by the presence of ≥ 1 Gadolinium (Gd)-enhancing T1 lesion in the screening MRI scan or by ≥ 4 new or enlarging T2 lesions in the screening scan as compared to a reference scan
* Participants who have active progressive multifocal leukoencephalopathy (PML), have had confirmed PML, or have a high degree of suspicion for PML
* Known presence of other neurological disorders that may mimic MS including but not limited to: neuromyelitis optica spectrum disease, Lyme disease, untreated Vitamin B12 deficiency, neurosarcoidosis, cerebrovascular disorders, and untreated hypothyroidism
* Known active or uncontrolled bacterial, viral, fungal, mycobacterial infection or other infection, excluding fungal infection of nail beds, including participants exhibiting symptoms consistent with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) within 6 weeks prior to Day 1
* Participants with a current diagnosis of epilepsy
* Clinically significant cardiac, metabolic, hematologic, hepatic, immunologic, urologic, endocrinologic, neurologic, pulmonary, psychiatric, dermatologic, allergic, renal, or other major diseases
* History of cancer, including hematologic malignancy and solid tumors, within 10 years of screening. Basal or squamous cell carcinoma of the skin that has been excised and is considered cured and in situ carcinoma of the cervix treated with apparent success by curative therapy >1 year prior to screening is not exclusionary
* Any concomitant disease that may require treatment with systemic corticosteroids or immunosuppressants during course of the study
* History of currently active primary or secondary (non-drug-related) immunodeficiency
* History of hypersensitivity to biologic agents or any of the excipients in the formulation
* Only for cohorts where CSF samples are planned to be collected: Participants with a history of spinal cord compression, raised intra-cerebral pressure, clinically significant vertebral joint pathology or any other current abnormalities in the lumbar region which could prevent the lumbar puncture procedure.

Prior/Concomitant Therapy:

* Treatment with any approved MS treatment at Screening. Participants may become eligible after completion of a washout period prior to acquiring any screening laboratory tests but should not be withdrawn from therapies for the sole purpose of meeting eligibility for the trial
* Previous treatment with RO7121932, alemtuzumab, cladribine, mitoxantrone, cyclophosphamide, total body irradiation, bone marrow transplantation, and hematopoietic stem cell transplantation. For the USA only, previous treatment with daclizumab
* Previous treatment with anti-cluster of differentiation 20 (CD20) B-cell-depleting therapies (e.g., rituximab, ocrelizumab, or ofatumumab)

  * <12 months prior to acquiring any screening laboratory tests,
  * ≥12 months prior to acquiring any screening laboratory tests, if B-cells are outside the normal range, or not back to individual baseline ± 20% (if data are available),
  * If discontinuation of a prior B-cell depletion therapy was motivated by safety reasons
* Current or prior treatment with natalizumab (if <24 months prior to acquiring any screening laboratory tests)

Prior/Concurrent Clinical Study Experience:

- Participation in an investigational drug medicinal product or medical device study within 30 days before Screening or within five times the pharmacodynamic (PD) or pharmacokinetic (PK) half-life (if known), whichever is longer

Diagnostic Assessments:

* Positive result on human immunodeficiency virus (HIV1) and HIV2, hepatitis C, or hepatitis B
* Participants with SI or behavior within 6 months prior to Screening or participants who, in the Investigator's judgment, pose a suicidal or homicidal risk
* Vaccination with a live or live-attenuated vaccine within 6 weeks prior to Day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2027-07-08 (Estimated); Study Completion 2027-07-08 (Estimated)

PRIMARY OUTCOMES:
Parts 1, 2, and 3: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) With Severity of AEs Measured According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5 (NCI CTCAE V5) | Day 1 to Day 169 for Part 1 and Part 2; Day 1 to Day 197 for Part 3
Parts 1, 2, and 3: Change From Baseline in Suicide Risk as Assessed Using the Columbia-Suicide Severity Rating Scale (C-SSRS) | Day 1 to Day 169 for Part 1 and Part 2; Day 1 to Day 197 for Part 3
  The C-SSRS is an interview-based instrument used to assess baseline incidence of suicidal ideation (SI) and behavior. The assessment includes "yes" or "no" responses for 5 questions, each related to SI (wish to be dead, non-specific active suicidal thoughts, active SI with any methods, active SI with some intent, active SI with specific plan) and suicidal behavior (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, suicide). Numeric ratings are provided for severity of ideation (if present), from 0 to 5. A score of 0 is assigned if no suicide risk is present. A score of 1 or higher indicates SI or behavior, with 5 being the most severe.
Parts 2 and 3: Percentage of Participants With Local Pain at the Site of Injection Assessed Using the Visual Analog Scale (VAS) | Day 1, 2, 5, 8 for Part 2; Day 1, 2, 5, 8, 15, 22, 29, 36 for Part 3
  VAS is a 100 millimetre (mm) horizontal visual analog scale with values 0 to 100 mm to indicate pain. The following cutpoints on the VAS will be considered in the interpretation of the pain data: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm). A higher score indicates greater pain intensity.
Parts 2 and 3: Percentage of Participants With Local Injection-site Reaction Using Local Injection-site Symptom Assessment (LISSA) | Day 1,2, 5, 8 for Part 2; Day 1, 2, 5, 8, 15, 22, 29, 36 for Part 3
  LISSA form will be used to assess the participant's injection site for the following categories of reactions: Burning, Itching, Bruising, Erythema (redness), Hive formation, Induration, Swelling, Ecchymosis, Sensitivity, Papules, Stinging, Blister, Cold sensation, and Other. These reactions will be described using the following scale: Unable to assess, less than a dime (<18 mm/<0.7 inches), a dime (18 mm/0.7 inches), a nickel (21 mm/0.8 inches), a quarter (24 mm/1 inch), a half dollar (31 mm/1.2 inches), larger than a half dollar (>31 mm/>1.2 inches). A higher score indicates high injection site reactions.

SECONDARY OUTCOMES:
Parts 1, 2 and 3 (Week 1 and Week 4): Time to Maximum Observed Concentration (Tmax) of RO7121932 | Day 1 to Day 169 for Part 1 and Part 2; Days 1, 2, 5 and, 22 for Part 3
Parts 1, 2 and 3 (Week 1 and Week 4): Maximum Observed Serum Concentration (Cmax) of RO7121932 | Day 1 to Day 169 for Part 1 and Part 2; Days 1, 2, 5 and, 22 for Part 3
Parts 1, 2 and 3 (Week 1 and Week 4): Area Under the Serum Concentration-time Curve From Time 0 to 168 Hours (h) (AUC0-168h) Postdose | Day 1 (predose) to Day 8 (168 hours post-dose) for Parts 1, 2, and 3 (Week 1) and Day 22 (predose) to Day 29 (168 hours post-dose) for Part 3 (Week 4)
Parts 1 and 2: Area Under the Serum Concentration-time Curve up to the Last Measurable Concentration (AUClast) | Day 1 to Day 169 for Part 1 and Part 2
Parts 1 and 2: AUC From Time 0 to Infinity (AUCinf) | Day 1 to Day 169 for Part 1 and Part 2
Part 1: Total Body Clearance (CL) Of RO7121932 | Day 1 to Day 169
Parts 2 and 3 (Week 4): Apparent Clearance (CL/F) of RO7121932 | Day 1 to Day 169 for Part 2; Day 22 to Day 29 for Part 3
Parts 1, 2 and 3: Terminal Rate Constant of RO7121932 | Day 1 to Day 169 for Part 1 and Part 2; Day 22 to Day 197 for Part 3
Parts 1, 2 and 3: Apparent Terminal Half-Life (T1/2) of RO7121932 | Day 1 to Day 169 for Part 1 and Part 2; Day 22 to Day 197 for Part 3
Part 3: Trough Concentrations (Ctrough) of RO7121932 | Day 1 to Day 197
Part 3 (Week 1 and Week 4): Area Under the Concentration-time Curve Over One Dosing Interval (AUCtau) of RO7121932 | Day 1, 2, 5 and 22
Parts 1 and 3: Cerebrospinal Fluid (CSF) Concentration of RO7121932 | Screening, Day 2 to Day 169 for Part 1; Screening, Day 2 to Day 197 for Part 3
Parts 1, 2, and 3: Percentage of Participants With Anti-RO7121932 Antibodies | Days 1, 8, 22, 29, 57, 85,169 for Part 1; Days 1, 8, 22, 57, 85, 169 for Part 2; Days 1, 8, 15, 22, 29, 57, 85, 120 & 197 for Part 3
Parts 1, 2, and 3: Time Course of B-cell Frequencies in Blood | Screening, Days 1, 2, 8, 22, 57, 85, 169 for Part 1; Screening, Days 1, 2, 8, 22, 57, 85, 169 for Part 2; Screening, Days 1, 2, 8, 15, 22, 57, 85, 120, 197 for Part 3
Part 1: Time Course of B-cell Frequencies in CSF | Screening, Day 2 to 169
Parts 1, 2, and 3: Change From Baseline in B-cell Frequencies in Blood | Screening, Days 1, 2, 8, 22, 57, 85, 169 for Part 1; Screening, Days 1, 2, 8, 22, 57, 85, 169 for Part 2; Screening, Days 1, 2, 8, 15, 22, 57, 85, 120, 197 for Part 3
Parts 1 and 3: Change From Baseline in B-cell Frequencies in CSF | Screening, Day 2 to 169 for Part 1; Screening, Day 2 to 197 for Part 3

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (32):
- United States (5):
  - Stanford University Medical Center, Stanford, California
  - Yale University Multiple Sclerosis Center, New Haven, Connecticut
  - University of South Florida, Tampa, Florida
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - UC Health, LLC., Cincinnati, Ohio
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Gent, Ghent
- Montreal Neurological Institute and Hospital, Montreal, Quebec, Canada
- Germany (6):
  - Universitätsklinikum "Carl Gustav Carus", Dresden
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
  - Klinikum rechts der Isar der TU Muenchen, München
  - Universitätsklinikum Münster Klinik u. Poliklinik f. Neurologie, Münster
  - Universitätsklinikum Tübingen, Zentrum für Neurologie, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Israel (2):
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Fond. Istituto Neurologico C.Besta, Milan, Lombardy
- ARENSIA Exploratory Medicine Phase I, PMSI Republican Clinical Hospital, Chisinau, Moldova
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Regionalny Szpital Specjalistyczny im. W. Bieganskiego, Grudzi?dz
  - MedPolonia, Poznan
  - Osrodek Badan Klinicznych Euromedis, Szczecin
  - Instytut Psychiatrii i Neurologii II Klinika Neurologiczna, Warsaw
  - SPSK nr 1, Zabrze
- Portugal (3):
  - Hospital de Braga, Braga
  - Hospital Santo Antonio dos Capuchos, Lisbon
  - Centro Hospitalar Entre o Douro e Vouga E.P.E. - Hospital de São Sebastião, Santa Maria da Feira
- Romania (2):
  - ARENSIA Exploratory Medicine SRL - Bucharest (Monza Medical Center), Bucharest
  - ARENSIA Exploratory Medicine, County Emergency Hospital, Cluj-Napoca
- University Clinical Center of Serbia, Belgrade, Serbia
- Hospital Universitari Vall dHebron (CEMCAT), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing